CLINICAL TRIAL: NCT07116733
Title: Desflurane vs. Propofol for Cardiac Anesthesia: Impact on Developing Major Cardiac Events in Patients Undergoing CABG Procedure
Brief Title: Desflurane vs. Propofol for Cardiac Anesthesia
Acronym: DECIDE-CABG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal investigator, Chief of Anesthesia Clinical Research Center, Xijing Hospitall, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20250104
Record Dates: First submitted 2025-08-06; First posted 2025-08-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Surgery; Coronary Artery Bypass Grafting
Keywords: Desflurane; Propofol; Cardiac Surgery; Major Cardiac Event; Coronary Artery Bypass Grafting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane group (Experimental): After routine induction, anesthesia is maintained with inhaled desflurane, with the concentration adjusted as needed to maintain 0.5-2 MAC .Propofol is not used to maintain anesthesia during the whole anesthesia maintenance process, except during cardiopulmonary bypass.
  Interventions: Drug: Desﬂurane group
- Propofol group (Active Comparator): 3-8 mg/kg/h intravenous infusion of propofol to implement total intravenous anesthesia maintenance, without the use of any inhaled anesthetic drugs, can be maintained by intravenous targeted infusion or manual adjustment of intravenous infusion.
  Interventions: Drug: Propofol group

INTERVENTIONS:
Drug: Desﬂurane group — After routine induction, maintain anesthesia with inhaled desflurane , adjusting concentration as needed to sustain 0.5-2 MAC . To maximize the cardioprotective effects of inhaled anesthetics, adhere to this intraoperative strategy:
  Maintain ≥1 MAC continuous desflurane for ≥30 minutes ; For on-pump CABG , discontinue desflurane 15 minutes before initiating cardiopulmonary bypass (CPB) ;
  If intraoperative desflurane cessation is required, implement a wash-in/wash-out strategy (recommended but non-mandatory):
  Perform 3 alternating cycles of:
  Wash-in : ≥10 minutes of desflurane at ≥0.5 MAC, Wash-out : ≥10 minutes of complete cessation of inhaled anesthetics. Propofol is strictly prohibited for anesthesia maintenance throughout the procedure , except during CPB.
  Arms: Desflurane group
Drug: Propofol group — Administer total intravenous anesthesia (TIVA) using propofol infusion at 3-8 mg/kg/h . No inhaled anesthetics are permitted for maintenance. This may be delivered via:target-controlled infusion (TCI) systems, or manual adjustment of intravenous infusion rates.
  Arms: Propofol group

SUMMARY:
To investigate whether the inhaled anesthetic desflurane, compared with propofol, exerts cardioprotective effects and reduces the incidence of severe postoperative major cardiac events in patients undergoing coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
Cardiac surgery is among the highest-risk surgical procedures, with a high incidence of severe postoperative complications that affect patient prognosis. It is a critical factor significantly increasing perioperative mortality and poses a major challenge to the prognosis of patients undergoing cardiac surgery. Coronary-artery bypass grafting (CABG) is the most common cardiac surgery, with over 300,000 procedures performed annually in the United States alone. The incidence of cardiac complications after cardiac surgery is as high as 50%, including approximately 35% for new-onset atrial fibrillation, 30% for acute kidney injury, 16% for respiratory failure, 5% for severe infection, and an in-hospital mortality rate of about 3.5%. Key pathogenic factors contributing to severe complications after cardiac surgery include surgical stress responses, insufficient organ perfusion during perioperative management, and tissue/organ damage or dysfunction caused by oxidative stress responses induced by the release of inflammatory factors.

Outcomes and prognosis following cardiac surgery are influenced by patient characteristics, surgical techniques, and perioperative management. Over the years, we have continuously sought to develop effective strategies to reduce the incidence of perioperative complications and mortality. Anesthesia for CABG (Coronary Artery Bypass Graft) is typically induced solely with intravenous agents (Total Intravenous Anesthesia - TIVA) or using a combination of volatile (inhaled) and intravenous agents. When administered prior to, during, or after an ischemic event, volatile anesthetics exert cytoprotective effects via multiple mechanisms. These include modulating G protein-coupled receptors, intracellular signaling pathways, gene expression, potassium channels, and mitochondrial function . Furthermore, volatile anesthetics reduce myocardial infarct size in animal models. Several randomized controlled trials (RCTs) suggest volatile anesthetics can reduce biomarkers of myocardial injury, even when administered for only a brief period before ischemia. Additionally, inhaled anesthetics , besides reducing postoperative cardiac troponin release and preserving cardiac function after cardiac surgery, may also lower the risk of myocardial infarction .

However, the impact of volatile anesthetics on postoperative complications and mortality following cardiac surgery remains inconsistent. Some meta-analyses have demonstrated reduced mortality after CABG with volatile anesthetics, a finding consistent with observations from moderate-sized randomized controlled trials. Two international consensus conferences identified volatile anesthetics as key non-surgical interventions to improve survival in patients undergoing major surgery, with potential significant clinical implications for over 300 million surgical patients annually. Guidelines from the American College of Cardiology, American Heart Association, and European Association for Cardio-Thoracic Surgery recommend applying these findings to anesthetic management in cardiac surgery patients, advocating inhalational anesthetics for maintenance in patients at cardiovascular risk to reduce postoperative complications. However, other randomized controlled trials and meta-analyses have failed to confirm such benefits. Conflicting results also exist regarding postoperative complications, including pulmonary complications, neurocognitive disorders, and renal injury.

The large-scale international multicenter Myriad trial-designed to enroll 10,600 patients undergoing isolated CABG to compare inhalational anesthetics (isoflurane, sevoflurane, or desflurane) versus intravenous propofol on postoperative mortality-the study was prematurely terminated for futility after enrolling 5,400 CABG cases. Interim analysis revealed no differences in 30-day and 1-year all-cause mortality between volatile anesthesia and total intravenous anesthesia (TIVA) groups. Another multicenter study (Br J Anaesth. 2024 Aug;133(2):296-304), involving 3,123 cardiac surgery patients across 16 Chinese centers, compared inhalational (sevoflurane/desflurane) and intravenous (propofol) anesthesia for composite outcomes including 30-day all-cause mortality and severe organ complications. No significant difference was observed: 33.8% in the inhalational group versus 33.2% in the intravenous group (adjusted OR 1.05, 95% CI 0.90-1.22; P=0.57).

Desflurane , introduced into clinical practice in 1990 as an inhaled anesthetic, is characterized by rapid induction and recovery , contributing to reduced postoperative recovery-related complications . Studies confirm that desflurane anesthesia lowers the surgical stress response , aiding in the maintenance of hemodynamic stability . Furthermore, multiple studies have found that compared to intravenous anesthesia, desflurane offers superior myocardial protection for CABG patients, reducing pulmonary complications, shortening hospital stays, lowering mortality, and improving quality of life . Its mechanisms may relate to its effects on mitochondrial permeability transition pore, mitochondrial electron transport chain, reactive oxygen species, ATP-sensitive potassium channels, G protein-coupled receptors, and protein kinase C biological functions. In non-cardiac surgery, desflurane did not reduce postoperative respiratory complications compared to sevoflurane . Although clinical evidence supporting the beneficial effects of inhaled anesthetics, particularly desflurane, in cardiac surgery patients is limited and insufficient , they do highlight its potential advantages . Research into desflurane's optimal administration method and dosage , as well as its long-term effects , is ongoing.

A recently published Meta-analysis indicated that, compared to propofol , desflurane demonstrated potential clinical benefit for surgical patients in terms of 30-day mortality, incidence of myocardial infarction, new-onset postoperative atrial fibrillation, postoperative pneumonia, and atelectasis . However, these findings stemmed from small sample sizes and underpowered studies .

Based on the available evidence, the inconsistent conclusions across current studies may stem from :

1. Differential organ-specific effects of inhalational versus intravenous anesthetics: Inhalational agents confer significant cardiovascular benefits, whereas intravenous agents offer neurological advantages. Consequently, using mortality or composite outcomes encompassing severe complications across all organ systems as primary endpoints leads to confounding of divergent effects, posing challenges for result interpretation and clinical practice guidance.
2. Heterogeneity in cardioprotective efficacy among inhalational agents: Existing studies have not restricted the type of inhalational anesthetics used. When compared to the intravenous agent propofol, commonly used inhalational anesthetics (isoflurane, desflurane, sevoflurane) exhibit heterogeneous cardioprotective effects: isoflurane shows weaker cardioprotection than propofol; sevoflurane demonstrates no significant difference; and desflurane exhibits stronger cardioprotection than propofol.
3. Impact of timing and duration of inhalational anesthetic administration: In clinical practice, the timing and duration of inhalational agent use influence their cardioprotective efficacy, representing a key source of effect heterogeneity across studies.

To date, no study has provided robust evidence supporting a preferred anesthesia regimen or agent for preventing severe complications and reducing mortality after cardiac surgery. Building upon the potential advantages of desflurane in myocardial protection and improving postoperative survival , identified in preliminary small-scale studies or exploratory analyses of other large trials , we plan to initiate a large-scale, national, multi-center randomized clinical trial (DECIDE-CABG trial) .

This trial will enroll 3,560 elective patients undergoing isolated CABG to compare the impact of desflurane-based inhaled anesthesia maintenance versus propofol-based TIVA maintenance on the incidence of major adverse cardiovascular events (MACE) and all-cause mortality at 30 days postoperatively . Through this large-scale, multi-center, randomized controlled study , we aim to definitively identify the optimal anesthesia regimen and anesthetic agents for CABG patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective coronary artery bypass grafting (CABG)
2. Age ≥ 18 years old;
3. Sign the informed consent form.

Exclusion Criteria:

1. Emergency or urgent operation
2. Concomitant valve or aortic surgery
3. History of myocardial infarction in recent 30 days
4. Current use of myocardial preconditioning-affecting medications, such as sulfonylurea (glibenclamide), allopurinol, theophylline, nicorandil(last dose < 8 hrs), etc
5. Participated in other randomized controlled clinical trials in recent 3 months
6. General anesthesia in recent 30 days
7. History of kidney and liver transplantation, or severe liver and kidney dysfunction (EGFR ≤ 20 mlgmin/1.73 m2, conventional dialysis or patients who have started dialysis; Child Pugh grade C/cirrhosis)
8. History of open heart surgery;
9. Hemodynamic instability or severe heart failure (SBP<90 mmHg or preoperative need of high-dose vasoactive drug support, placement of aortic balloon pump (IABP), ECMO or ventricular assist device, left ventricular ejection fraction<30%)
10. Adverse drug reactions to trial medications
11. History of malignant hyperthermia
12. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3560 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of death and major cardiac events | within 30 days after operation
  It is composite outcome including:
  1. All-cause mortality within 30 days postoperatively
  2. New-onset acute heart failure, or any of the following: Cardiac arrest with successful resuscitation; Cardiogenic shock requiring mechanical circulatory support: Intra-aortic balloon pump (IABP), Extracorporeal membrane oxygenation (ECMO), Left ventricular assist device (e.g., Impella); Low cardiac output syndrome necessitating high-dose inotropic support (Inotropic Score (IS) >15 within the first 24 postoperative hours, IS >10 within 48 postoperative hours).
  3. Arrhythmia requiring intervention: New-onset atrial fibrillation (pharmacotherapy or pacemaker),Other clinically significant arrhythmias.
  4. Acute myocardial infarction
  5. Emergency sternotomy/re-exploration for: Cardiac tamponade, Uncontrolled hemorrhage, Other life-threatening complications.

SECONDARY OUTCOMES:
Incidence of death and the major cardiac events | within 30 days after operation
  the incidence of each component outcome in the primary outcome
Total number of death and major cardiac events | within 30 days after operation
  Total number of events listed as the components of the primary outcomes.
Length of mechanical ventilation | within 30 days after operation
  Length of mechanical ventilation in hours
Length of lCU stay | From the date of surgery until the date patient discharge from hospital, assessed up to 1 year
  Length of postoperative lCU stay
Incidence of pulmonary complications | within 30 days after operation
  Including pulmonary infection, pleural effusion, respiratory failure, acute respiratory distress syndrome, pneumothorax, pulmonary embolism
Incidence of renal complications | within 30 days after operation
  Including AKI and RRT
Incidence of neurological complications | within 30 days after operation
  Including delirium, stroke, cognitive impairment
Readmission | within 30 days after operation
  Readmission after hospital discharge
All cause 90 d mortality | within 90 davs after operation
  Death within 90 days after surgery for any reason

OTHER OUTCOMES:
SOFA score | during postoperative ICU stay, with an average of 10 days
  Daily SOFA scores during ICU stay
The need for blood product transfusions | from the day of surgery to hospital discharge, average for 7-10 days
  The volume of RBCs, Platelet, FFP transfusion
Volume of chest tube drainage | within 72 hours following surgery
Requirement for vasoactive agents support for more than 48 hours | at 48 hours following surgery
The maximum VIS (Vasoactive-Inotropes Score) | within 7 days following surgery
incidence of postoperative infection | from end of surgery until hospital discharge, average for 10 days
  including pneumonia, deep sternal wound infection/mediastinitis, endocarditis, central venous catheter-related infection, urinary tract infection
the Kansas City Cardiomyopathy Questionnaire (KCCQ) | at 90 days and 1 years following surgery
  KCCQ measures symptoms, physical and social limitations, and quality of life in patients with heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, M.D., phd, Principal Investigator — Xijing Hospital
Locations (14):
- China (14):
  - Fuzhou University Affiliated Provincial Hospital, Fuzhou, Fujian
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjin, Jiangsu
  - Xijing Hospital, Xi'an, Shaanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - Daping Hospital, Army Medical University, Chongqing
  - Changhai Hospital, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
The sharing ofindividual Patient Data (lPD) will be considered at 1 year after the publication ofthe primary resultsf the project. Any request for lPD sharing Investigator (Pl), clearly outlining the intended use of the data.should be submitted as a proposal to the Pl, clearly outlining the intended use of the data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: beginning 12 morths after publication of the primary results
Access Criteria: Investigators who provide a methodologically sound proposal and whose proposed use of data has been approved by the steering committee. For instance for using lPD data for meta- analysis. Proposals sholId be submitted to principle investigator and committee the trial. To gain access, data requestors will need to sign a data access agreement

REFERENCES:
- [Background] Kampman JM, Hermanides J, Hollmann MW, Gilhuis CN, Bloem WA, Schraag S, Pradelli L, Repping S, Sperna Weiland NH. Mortality and morbidity after total intravenous anaesthesia versus inhalational anaesthesia: a systematic review and meta-analysis. EClinicalMedicine. 2024 May 14;72:102636. doi: 10.1016/j.eclinm.2024.102636. eCollection 2024 Jun. PMID 38774674
- [Background] Qin H, Zhou J. Myocardial Protection by Desflurane: From Basic Mechanisms to Clinical Applications. J Cardiovasc Pharmacol. 2023 Sep 1;82(3):169-179. doi: 10.1097/FJC.0000000000001448. PMID 37405905
- [Background] Zangrillo A, Lomivorotov VV, Pasyuga VV, Belletti A, Gazivoda G, Monaco F, Nigro Neto C, Likhvantsev VV, Bradic N, Lozovskiy A, Lei C, Bukamal NAR, Silva FS, Bautin AE, Ma J, Yong CY, Carollo C, Kunstyr J, Wang CY, Grigoryev EV, Riha H, Wang C, El-Tahan MR, Scandroglio AM, Mansor M, Lembo R, Ponomarev DN, Bezerra FJL, Ruggeri L, Chernyavskiy AM, Xu J, Tarasov DG, Navalesi P, Yavorovskiy A, Bove T, Kuzovlev A, Hajjar LA, Landoni G; MYRIAD Study Group. Effect of Volatile Anesthetics on Myocardial Infarction After Coronary Artery Surgery: A Post Hoc Analysis of a Randomized Trial. J Cardiothorac Vasc Anesth. 2022 Aug;36(8 Pt A):2454-2462. doi: 10.1053/j.jvca.2022.01.001. Epub 2022 Jan 7. PMID 35168907
- [Background] Landoni G, Lomivorotov VV, Nigro Neto C, Monaco F, Pasyuga VV, Bradic N, Lembo R, Gazivoda G, Likhvantsev VV, Lei C, Lozovskiy A, Di Tomasso N, Bukamal NAR, Silva FS, Bautin AE, Ma J, Crivellari M, Farag AMGA, Uvaliev NS, Carollo C, Pieri M, Kunstyr J, Wang CY, Belletti A, Hajjar LA, Grigoryev EV, Agro FE, Riha H, El-Tahan MR, Scandroglio AM, Elnakera AM, Baiocchi M, Navalesi P, Shmyrev VA, Severi L, Hegazy MA, Crescenzi G, Ponomarev DN, Brazzi L, Arnoni R, Tarasov DG, Jovic M, Calabro MG, Bove T, Bellomo R, Zangrillo A; MYRIAD Study Group. Volatile Anesthetics versus Total Intravenous Anesthesia for Cardiac Surgery. N Engl J Med. 2019 Mar 28;380(13):1214-1225. doi: 10.1056/NEJMoa1816476. Epub 2019 Mar 19. PMID 30888743
- [Background] Han J, Ryu JH, Jeon YT, Koo CH. Comparison of Volatile Anesthetics Versus Propofol on Postoperative Cognitive Function After Cardiac Surgery: A Systematic Review and Meta-analysis. J Cardiothorac Vasc Anesth. 2024 Jan;38(1):141-147. doi: 10.1053/j.jvca.2023.09.038. Epub 2023 Oct 2. PMID 37919165
- [Background] Jiang JL, Zhang L, He LL, Yu H, Li XF, Dai SH, Yu H. Volatile Versus Total Intravenous Anesthesia on Postoperative Delirium in Adult Patients Undergoing Cardiac Valve Surgery: A Randomized Clinical Trial. Anesth Analg. 2023 Jan 1;136(1):60-69. doi: 10.1213/ANE.0000000000006257. Epub 2022 Oct 27. PMID 36301724
- [Background] Bonanni A, Signori A, Alicino C, Mannucci I, Grasso MA, Martinelli L, Deferrari G. Volatile Anesthetics versus Propofol for Cardiac Surgery with Cardiopulmonary Bypass: Meta-analysis of Randomized Trials. Anesthesiology. 2020 Jun;132(6):1429-1446. doi: 10.1097/ALN.0000000000003236. PMID 32205551
- [Background] Sousa-Uva M, Neumann FJ, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur J Cardiothorac Surg. 2019 Jan 1;55(1):4-90. doi: 10.1093/ejcts/ezy289. No abstract available. PMID 30165632